CLINICAL TRIAL: NCT04789317
Title: Pullback Pressure Gradient (PPG) Global Registry: Prospective Evaluation of the Impact of the PPG Index on Clinical Decision Making and Outcomes
Brief Title: Pullback Pressure Gradient (PPG) Global Registry
Acronym: PPG Global
Status: Active, not recruiting | Type: Observational
Sponsor: VZW Cardiovascular Research Center Aalst (Other)
Responsible Party: Sponsor
Other Study IDs: CRI050
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Chronic Coronary Insufficiency; Non ST Elevation Myocardial Infarction
Keywords: FFR; PPG; PCI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stable CAD or stabilized NSTEMI (ACS) with significant epicardial lesions defined as FFR≤0.80.: The PPG Global Registry an investigator-initiated, observational, multicenter study of patients with an indication for PCI based on coronary angiography and FFR ≤0.80. After confirmation of intention to treat with PCI, a manual pullback with PPG analysis will be performed. A second level of decision making is then performed concerning PCI, coronary artery bypass grafting (CABG) or medical therapy (OMT). Patients will undergo PCI at operator discretion and post-PCI FFR will be measured. Clinical follow-up will be performed at 1, 2 and 3 years.

SUMMARY:
The purpose of this study is to determine the predictive capacity of the Pullback Pressure Gradient (PPG) index for post-PCI FFR and to determine the impact of the PPG index on clinical decision making about revascularization and on clinical outcomes.

DETAILED DESCRIPTION:
A Fractional Flow Reserve (FFR) evaluation comprises measurement of a distal single value and a pullback maneuver during hyperemic conditions. The PPGindex is a novel metric derived from the FFR pullback curve.3 This metric complements the distal FFR value by informing the spatial distribution of epicardial resistance (i.e. focal or diffuse) along the coronary vessel. The PPGindex relies on two components: first, the magnitude of pressure drop determined as a maximal pressure gradient over 20 millimeters relative to the total vessel gradient; and second, the length of functional disease relative to total vessel length. These two parameters are weighted equally to provide a metric that ranges from 0 to 1. PPGindex values approaching 1 represent functional focal coronary artery disease (CAD) whereas values close to 0 represent diffuse functional CAD. Until now, the interpretation of the FFR pullback relied on visual assessment. The PPGindex quantifies the pattern of functional CAD and has been shown to predict functionally complete revascularization. Percutaneous revascularization in vessels with high PPGindex is associated with high post-PCI FFR and vast improvement in epicardial conductance whilst PCI in vessels with low PPGindex results in low post-PCI FFR. An curvilinear relationship is observed between PPGindex and functional gain (i.e. FFR post-PCI minus FFR pre-PCI). The PPGindex, therefore, aims to predict the response to PCI in physiological terms.

Calculation of the PPGindex is indicated in cases with an FFR≤0.80. FFR pullbacks are performed under hyperemic conditions at a steady pace during manual pullback. A calculation of the PPGindex using the Coroflow console (Coroventis Research Ab, Uppsala, Sweden) is available for online use and computes the PPG value immediately after the pullback maneuver. This software also includes an automated drift correction. The pullback curve is depicted on an dedicated pullback display screen and the pressure gradients are shown per millimeter, allowing correlation between the location of pressure step-ups and the anatomical target for PCI. In summary, we can distinguish three points where FFR influences the clinical decision-making process. First, an FFR ≤0.80 indicates potential benefit of revascularization. Second, the pullback curve assesses disease pattern and PPG index value quantifies it, helping de physician in the decision about treatment options (e.g. PCI, CABG or OMT). And, third, the location of pressure step-ups along the vessels helps plan the PCI strategy with respect to coverage of functional disease. A combined FFR and PPG-guided PCI strategy has the potential to improve patient selection and enhance procedural planning.

The purpose of this study is to determine the predictive capacity of the PPG index for post-PCI FFR and to determine the impact of the PPG index on clinical decision making about revascularization and on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with stable coronary artery disease or stabilized acute coronary syndrome and invasive FFR measurement ≤0.80.

Exclusion Criteria:

* Angiographic exclusion criteria

  1. Ostial lesions.
  2. Severe vessel tortuosity.
  3. Vessel rewiring deemed 'difficult' by the operator.
  4. Bifurcation with planned two-stent strategy.
  5. NSTEMI culprit vessel.
  6. STEMI
  7. Uncontrolled or recurrent ventricular tachycardia.
  8. Hemodynamic instability
  9. Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with stable coronary artery disease or stabilized acute coronary syndrome and indication for hemodynamic assessment by FFR and subsequent confirmation of significant epicardial CAD assessed by an invasive FFR measurement ≤0.80.
Sampling Method: Non-Probability Sample
Enrollment: 982 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive capacity of the PPG index for post-PCI FFR. | 1 year
  Describe the relationship between pre PCI PPG and post-PCI FFR

SECONDARY OUTCOMES:
To assess the relationship between baseline PPG index and major adverse cardiovascular events (cardiac death, peri-procedural and spontaneous myocardial infarction and target vessel revascularization) at one, two and three years. | 3 years after completion of inclusion
  Assess whether the PPG and identification of CAD endo-type has a relationship with per and post-procedure events
Difference between baseline and 12 month follow-up in the Seattle Angina Questionnaire (SAQ) stratified by PPG index. | 1 years after completion of inclusion
  Assess the relationship with symptoms assessed by the SAQ and PPG and persistent/recurrent angina post-PCI

OTHER OUTCOMES:
Rate of patients with intended PCI but deferred after PPG calculation. | 1 year
  Assess the influence of pullback and PPG on identification of patterns of CAD and change in treatment strategy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Collet, MD PhD, Principal Investigator — OLV Hospital
Locations (23):
- United States (3):
  - Stanford University, Stanford, California
  - St Francis Hospital and Heart Center, New York, New York
  - Memorial Hermann Texas Medical Center, Texas City, Texas
- Australia (2):
  - Monash Medical Center, Melbourne
  - Concord Repatriation General Hospital, Sydney
- OLV Aalst, Aalst, Belgium
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Righospitalet, Copenhagen
- Institut Arnault Tzanck, Nice, France
- Italy (2):
  - Ferrara University, Ferrara
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
- Japan (4):
  - Aichi University, Aichi
  - Gifu Heart Center, Gifu
  - Showa University Hospital, Tokyo
  - Tokyo D Tower Hospital, Tokyo
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Radboud UMC, Nijmegen
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Princesa, Madrid
- Karolinska Institutet, Stockholm, Sweden
- CHUV, Lausanne, Switzerland
- Guy and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collet C, Sonck J, Vandeloo B, Mizukami T, Roosens B, Lochy S, Argacha JF, Schoors D, Colaiori I, Di Gioia G, Kodeboina M, Suzuki H, Van 't Veer M, Bartunek J, Barbato E, Cosyns B, De Bruyne B. Measurement of Hyperemic Pullback Pressure Gradients to Characterize Patterns of Coronary Atherosclerosis. J Am Coll Cardiol. 2019 Oct 8;74(14):1772-1784. doi: 10.1016/j.jacc.2019.07.072. PMID 31582137
- [Derived] Hada M, Mizukami T, Ikeda K, Munhoz D, Brouwers S, Sonck J, Matsuo H, Shinke T, Ando H, Ko B, Biscaglia S, Rivero F, Engstrom T, Arslani K, Leone AM, Galante D, van Nunen LX, Fearon WF, Christiansen EH, Fournier S, Desta L, Yong A, Adjedj J, Escaned J, Nakayama M, Eftekhari A, Zimmermann FM, Sakai K, Storozhenko T, da Costa BR, Campo G, Berry C, Collison D, Johnson T, Amano T, Perera D, Jeremias A, Ali Z, De Bruyne B, Barbato P, Corradetti S, Stalikas N, Kechichian A, Bouisset F, Kakuta T, Johnson NP, Collet C. Impact of Sex on Residual Angina After Percutaneous Coronary Interventions. Catheter Cardiovasc Interv. 2025 Dec 17. doi: 10.1002/ccd.70419. Online ahead of print. PMID 41408672
- [Derived] Collet C, Munhoz D, Mizukami T, Sonck J, Matsuo H, Shinke T, Ando H, Ko B, Biscaglia S, Rivero F, Engstrom T, Arslani K, Leone AM, van Nunen LX, Fearon WF, Christiansen EH, Fournier S, Desta L, Yong A, Adjedj J, Escaned J, Nakayama M, Eftekhari A, Zimmermann FM, Sakai K, Storozhenko T, da Costa BR, Campo G, West NEJ, De Potter T, Heggermont W, Buytaert D, Bartunek J, Berry C, Collison D, Johnson T, Amano T, Perera D, Jeremias A, Ali Z, Pijls NHJ, De Bruyne B, Johnson NP. Influence of Pathophysiologic Patterns of Coronary Artery Disease on Immediate Percutaneous Coronary Intervention Outcomes. Circulation. 2024 Aug 20;150(8):586-597. doi: 10.1161/CIRCULATIONAHA.124.069450. Epub 2024 May 14. PMID 38742491
- [Derived] Munhoz D, Collet C, Mizukami T, Yong A, Leone AM, Eftekhari A, Ko B, da Costa BR, Berry C, Collison D, Perera D, Christiansen EH, Rivero F, Zimmermann FM, Ando H, Matsuo H, Nakayama M, Escaned J, Sonck J, Sakai K, Adjedj J, Desta L, van Nunen LX, West NEJ, Fournier S, Storozhenko T, Amano T, Engstrom T, Johnson T, Shinke T, Biscaglia S, Fearon WF, Ali Z, De Bruyne B, Johnson NP. Rationale and design of the pullback pressure gradient (PPG) global registry. Am Heart J. 2023 Nov;265:170-179. doi: 10.1016/j.ahj.2023.07.016. Epub 2023 Aug 21. PMID 37611857
- [Derived] Achim A, Johnson NP, Liblik K, Burckhardt A, Krivoshei L, Leibundgut G. Coronary steal: how many thieves are out there? Eur Heart J. 2023 Aug 7;44(30):2805-2814. doi: 10.1093/eurheartj/ehad327. PMID 37264699